CLINICAL TRIAL: NCT04667962
Title: Impact of the Change in Hospital Service of Caregivers During COVID-19 Health Crisis on Operational Strain
Acronym: CovIdeDocS
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-33; 2020-A02932-37 (Other: IDRCB)
Record Dates: First submitted 2020-12-13; First posted 2020-12-16 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Burnout, Caregiver
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital service change: This group is composed of caregivers who changed hospital service during COVID-19 health crisis.
  Interventions: Other: Online questionnaire
- No hospital service change: This group is composed of caregivers who have not changed hospital service during COVID-19 health crisis.
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire — Participants will have to complete 3 online self-questionnaires: the first one at enrollment, the second one 1 month after enrollment (M1) and the third one 3 months after enrollment (M3). Each questionnaire will take an estimated 20 minutes to complete.

SUMMARY:
The French Armed Forces Health Service caregivers are confronted with specific operational constraints that require physiological adaptation on a daily basis. These constraints generate an allostatic load resulting from the body's adaptation to the environment through stress response systems. The COVID-19 health crisis has modified the physical and psychological constraints linked to usual activity, in particular by imposing versatility to caregivers.

The research hypothesis is that carers who have undergone activity reorganisations, and in particular a change of service, are more affected by the health crisis than those who have remained in their service and have continued an activity close to their usual practice.

ELIGIBILITY:
Inclusion Criteria:

* To be caregivers
* Have been in employment between March 15 and May 15, 2020

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is composed of caregivers from the French Armed Forces Health Service (Medical doctor, nurse, assistant nurse, ...) who have been in employment when the COVID-19 health crisis began in France.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Burn-out Assessment tool (BAT) score at enrollment. | At enrollment
  Burn-out Assessment tool (BAT) score at enrollment will be compared between the "hospital service change" group and the "no hospital service change" group.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge
  - Ecole du Val-de-Grâce, Paris

IPD SHARING:
Plan to Share IPD: Undecided